CLINICAL TRIAL: NCT01878604
Title: The Study of Gene Analysis and Treatment Optimization in Chinese Homozygous Familial Hypercholesterolemia
Brief Title: Gene Analysis and Treatment Optimization in Chinese Homozygous Familial Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Shuiping Zhao, Chief of Cardiology Department, 2nd Xiangya Hospital, Central South University
Other Study IDs: MISP50469
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Homozygous Familial Hypercholesterolemia: Gene Analysis for Homozygous Familial Hypercholesterolemia cases
  Interventions: Genetic: Gene analysis; Other: Historical data of lipid-lowering drug administration; Other: Historical data of plasma lipids, xanthoma changes

INTERVENTIONS:
Genetic: Gene analysis — Gene analysis
Other: Historical data of lipid-lowering drug administration — Collecting historical data of lipid-lowering drug administration
Other: Historical data of plasma lipids, xanthoma changes — Collecting historical data of plasma lipids and xanthoma changes

SUMMARY:
Identify new or novel genes which may impact on cholesterol level, and establish the relationship between those gene mutations with atherosclerosis, as well as responses to lipid-lowering drugs.

DETAILED DESCRIPTION:
To better understand the genetics basis for LDL-C elevation and develop an optimized lipid-lowering strategy, we propose to do the following studies:

1. To establish a China HoFH registry, and collect DNA and blood samples from all available family members of each proband (pedigrees);
2. To detect gene mutations known to cause FH and identify family suitable for future whole genome sequencing aimed to identify novel genes controlling cholesterol levels.

3.To establish the relationship between types of gene mutations and lipid and atherosclerosis profile, as well as responses to lipid-lowering agents.

ELIGIBILITY:
Inclusion criteria:

Patients of any age and sex who meet clinical or genetic criteria for hoFH as follows:

* Cutaneous xanthomata before the age of ten years
* LDLC > 13 mmol/L before treatment or > 7.76 mmol/L despite treatment
* Phenotypic features in keeping with HeFH in both parents

Exclusion criteria:

Inability of patient, or, if less than 18, a parent, to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Homozygous Familial Hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2001-10; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuiping Zhao, Doctor, Principal Investigator — Central South University
Locations (1):
- Cardiology department of 2nd Xiangya Hospital, Changsha, Hunan, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homozygous Familial Hypercholesterolemia
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients of HoFH: patients of Homozygous Familial Hypercholesterolemia
Arm/Group | Patients of HoFH
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: year] | 5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
plasma LDL cholesterol concentration [Mean (Standard Deviation); unit: mmol/L] | 17.55 (2.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of LDLR Gene Mutations
Description: Number of gene mutations based on the sequencing results in terms of some known genes and suspected novel genes.
  c.796 G>C and c.1048 C>T in the LDLR gene c.1448 G>A and c.1720C>A in the LDLR gene c.2030 G >A and c.1257 C>A in the LDLR gene homozygous mutation c.605 T>C in the LDLR gene
Time Frame: 1 year
Measure: Number; unit: gene mutations
Groups:
- HoFH Patients: HoFH patients
Arm/Group | HoFH Patients
Number analyzed (Participants) | 5
gene mutations | 7

2. Secondary Outcome: LDL-C Reduction Percentage
Description: plasma LDL-C reduction percentage with lipid-lowering drugs from pre-treatment to the last time follow-up time point
  plasma LDL-C reduction percentage calculation: "plasma LDL-C at pre-treatment time point" minus "plasma LDL-C at the last time follow-up time point", and then compared with "plasma LDL-C at pre-treatment time point", namely "plasma LDL-C reduction percentage".
Time Frame: pre-treatment and 6-13 years post treatment
Measure: Mean (Standard Error); unit: percentage of plasma LDL-C reduction
Groups:
- HoFH Patients: patients of Homozygous Familial Hypercholesterolemia that meet the Inclusion criteria:
  * Cutaneous xanthomata before the age of ten years
  * LDLC > 13 mmol/L before treatment or > 7.76 mmol/L despite treatment
  * Phenotypic features in keeping with HeFH in both parents
Arm/Group | HoFH Patients
Number analyzed (Participants) | 5
percentage of plasma LDL-C reduction | 48.16 (8.5981)

ADVERSE EVENTS:
Description: Only serious adverse events were collected/assessed.
Groups:
- HoFH Patients: all HoFH patients enrolled in this study
Arm/Group | HoFH Patients
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No